CLINICAL TRIAL: NCT06045260
Title: "Receptor Radionuclide Therapy With 177Lu-DOTATOC (177Lu-edotreotide or 177Lu-octreotide) in SSTR Positive Patients: a Multicenter, Prospective, Phase II Trial"
Brief Title: "Receptor Radionuclide Therapy With 177Lu-DOTATOC
Acronym: LUFOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST 100.60
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Neuroendocrine Tumors; Paraganglioma; Pheochromocytoma
MeSH Terms: conditions — Neuroendocrine Tumors; Paraganglioma; Pheochromocytoma | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7.4 Gbq Dose (Experimental): Patients with less than 2 risk factors out of the following will receive a dose equal to 7.4 GBq of the experimental radiopharmaceutical 177Lutetium-DOTATOC:
  * Pre-existing renal impairment (Creatinine > 1.5 mg/dl and/or eGFR or creatinine clearance >50 and < 60 ml/min) or(chemotherapy, local external radiotherapy);
  * Patients who have received earlier nephrotoxic treatment modalities (chemotherapy, local external field radiation);
  * Relevant renal morphological abnormalities;
  * Previously major (G3-4) iatrogenic toxicities;
  * ECOG = 2;
  * Any previous Peptide Receptor Radionuclide Therapy;
  * Type 1 or 2 diabetes not controlled with therapy;
  * Arterial hypertension not controlled with therapy;
  * Extension of disease = 4 according to "tumor burden Krenning scale" (9);
  * Age (>80 years).
  Interventions: Drug: 177Lu-DOTATOC
- 5.5 Gbq Dose (Experimental): Patients with al least 2 risk factors out of the following will receive a dose equal to 5.5 GBq of the experimental radiopharmaceutical 177Lutetium-DOTATOC:
  * Pre-existing renal impairment (Creatinine > 1.5 mg/dl and/or eGFR or creatinine clearance >50 and < 60 ml/min) or(chemotherapy, local external radiotherapy);
  * Patients who have received earlier nephrotoxic treatment modalities (chemotherapy, local external field radiation);
  * Relevant renal morphological abnormalities;
  * Previously major (G3-4) iatrogenic toxicities;
  * ECOG = 2;
  * Any previous Peptide Receptor Radionuclide Therapy;
  * Type 1 or 2 diabetes not controlled with therapy;
  * Arterial hypertension not controlled with therapy;
  * Extension of disease = 4 according to "tumor burden Krenning scale" (9);
  * Age (>80 years).
  Interventions: Drug: 177Lu-DOTATOC

INTERVENTIONS:
Drug: 177Lu-DOTATOC — Administration of 4 cycles of therapy with 7.4 Gbq Dose for No risk factors Arm and 5.5 Gbq Dose for Risk Factor Arm. Both through slow intravenous infusion in 30 minutes with a dedicated pump system.

SUMMARY:
Peptide receptor radionuclide therapy (PRRT) may be recommended in G1- G2 GEP-NET patients with disease progression on somatostatine analogues therapy (LUTATHERA®). However, there are several diseases, including neuroendocrine neoplasia not originating from the digestive tract, for which the efficacy of PRRT has already been demonstrated, but which are not currently within the indications of LUTATHERA and therefore cannot benefit from it (i.e. bronchopulmonary, ovarian, renal NETs and neuroendocrine carcinomas). Moreover, the role of PRRT is also accepted in Pheochromocytomas and paragangliomas (PPGLs), Meningiomas, but also as a salvage therapy in pre-treated NET pts, and other SSTR-positive malignancies (Lymphomas, Gliomas…). Least explored among radiopharmaceuticals for SSTR-positive tumors is 177Lu-DOTATOC. This study aims to investigate the efficacy and safety of lutetium (177Lu) edotreotide (Lu-Dotatoc) on all the above-mentioned diseases that could benefit from receptor radionuclide therapy. We believe that this study, which will involve only patients outside the indication of LUTATHERA, will expand the current knowledge of radionuclide receptor therapy with 177Lu- DOTATOC, particularly with regard to objective response and safety parameters, and may consolidate its in the management of these diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients must have histologically or cytologically confirmation of neuroendocrine tumors or any other tumor histology type documented as sst2-positive, that may benefit from receptor radionuclide therapy and for which there are not any other effective treatments, included locoregional methods of control for PPGLs/pheochromocytoma. For cerebral and PPGLs sst2- positive tumors, if biopsy is no feasible for technical reason or risk benefit balance, patients may be enrolled if CT or MRI strongly suggest oncological lesion confirming the 68Ga PET-CT dota-peptide SSTr2 positivity.
3. Measurable disease according to RECIST 1.1 criteria also patients without measurable but with evaluable disease can be enrolled.
4. Any disease stage is allowed. Patients with documented disease will be admitted to the therapeutic phase only if the diagnostic PET/CT 68Ga-peptide images demonstrate a significant uptake in the tumour, according to the adapted Krenning Scale. Only patients with a greater caption (Grade 3 or 4) in most of the lesions will be admitted.
5. Patients with progressive disease in pre-study period (PD within the last 12 months), refractory to conventional standard treatments; clinical progression is allowed.
6. Patients with or without concurrent therapy with somatostatin analogs. It will be maintained the same dose of the SSA analogs as at the time of demonstrated disease progression.
7. Life expectancy of greater than 6 months.
8. ECOG performance status <2.
9. Adequate haematological, liver and renal function: haemoglobin >= 9 g/dL, absolute neutrophil count (ANC) >= 1.5 x 109 /L, platelets >= 100 x 109 /L, bilirubin ≤1.5 X UNL (upper normal limit), ALT and AST <2.5 X UNL (< 5 X UNL in presence of liver metastases), creatinine < 2 mg/dL and/or eGFR or creatinine clearance > 50 ml/min.
10. If female of childbearing potential highly effective birth control methods, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials", (2014_09_15 section 4.1) are mandatory (see Appendix F). Highly effective birth control methods are required beginning at the screening visit and continuing until 6 months following last treatment with study drug. A negative serum pregnancy test should be performed the same day the treatment is started at any cycle. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 6 months after final study drug administration. Two acceptable methods of birth control thus include Condom (barrier method of contraception) and one of the following is required (established use of oral, or injected or implanted hormonal method of contraception by the female partner; placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner; additional barrier method like occlusive cap with spermicidal foam/gel/film/cream/suppository in the female partner; tubal ligation in the female partner; vasectomy or other procedure resulting in infertility (eg, bilateral orchiectomy), for more than 6 months (see Appendix F).
11. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Patients treated with chemotherapy and therapeutic radiotherapy within 4 weeks and treated within 2 weeks with palliative radiotherapy, hormonal or biological therapy.
2. Known hypersensitivity to lutetium-177 (177Lu), edotreotide, DOTA or components of the formulation or other radiolabeled peptide agents.
3. Known hypersensitivity to lysine, arginine, or any excipient of the nephroprotective aminoacids given concurrently with the lutetium (177Lu) edotreotide infusion;
4. Patients treated with prior external beam radiation therapy (EBRT) to more than 25% of the bone marrow.
5. Patients treated with previous PRRT with an absorbed dose to the kidney more than 23 Gy and more than 1.8 Gy for the bone marrow or as surrogate of dosimetry (13).
6. Patients which are included in the indication of LUTATHERA®(9).
7. All acute toxic effects of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to a grade ≤ 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE).
8. ECOG performance status >2.
9. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Pregnant or breastfeeding women are excluded from the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy as Disease control rate (DCR) | 32 months
  percentage of patients who have achieved complete response, partial response, stable disease (according to RECIST 1.1) at the 1st planned evaluation.

SECONDARY OUTCOMES:
(Safety) percentage of patients who experience acute toxicity | 37 months
  evaluated according to version 5.0 CTC-AE (Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE). Safety is defined as the percentage of patients who experience acute toxicity from the 1st treatment until 30 days after the last treatment cycle or late toxicity that occurred after 30 days from the last treatment administration up to 6 months.
Progression free survival | 44 months
  Time from the start treatment date to the date of first observation of documented disease progression or death due to any cause.
Overall survival | 44 months
  Time from the therapy start to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.
Quality of life | 32 months
  Evaluated through validated standardized data collection forms from the EORTC QLQ-C30 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Sansovini, Study Chair — IRCCS IRST; Federica Matteucci, Principal Investigator — IRCCS IRST
Locations (2):
- Italy (2):
  - AUSL Romagna - Ospedale "M. Bufalini", Cesena, Forlì-Cesena
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l., Meldola, Forlì-Cesena